CLINICAL TRIAL: NCT02280785
Title: A Phase II Study of Brentuximab Vedotin for Relapsed/Refractory CD30-positive Non-Hodgkin Lymphomas Other Than Anaplastic Large Cell Lymphoma
Brief Title: Brentuximab Vedotin for Relapsed/Refractory CD30-positive Non-Hodgkin Lymphomas
Acronym: BRAN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Won Seog Kim, A phase II study of Brentuximab Vedotin for relapsed/refractory CD30-positive non-Hodgkin lymphomas other than anaplastic large cell lymphoma, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMC 2014-04-059
Record Dates: First submitted 2014-10-05; First posted 2014-11-03 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Brentuximab vedotin (Experimental): Brentuximab vedotin administered in 250ml of 0.9% saline by intravenous infusion over 30 minutes once every 3 weeks.
  In the absence of infusion toxicities, the infusion rate for all patients must be calculated in order to achieve a 30-minute (approximate) infusion period.
  Brentuximab Vedotin is dosed at 1.8mg/kg (capped at 100kg of body weight). Dosing is based on patients' weight according to the institutional standard; however, doses will be adjusted for patients who experience a ≥ 10% change in weight from baseline. Actual weight will be used except for patients weighing greater than 100 kg; dose will be calculated based on 100 kg for these individuals. The dose will be rounded to the nearest whole number of milligrams.
  Interventions: Drug: Brentuximab vedotin

INTERVENTIONS:
Drug: Brentuximab vedotin — Brentuximab vedotin must not be administered as an IV push or bolus. It must be administered in 100ml-250ml of 0.9% saline by intravenous infusion over 30 minutes once every 3 weeks.
  Other Names: Adcetris

SUMMARY:
Brentuximab vedotin is an antibody-drug conjugate targeting CD30, one of surface antigens expressed in lymphoma cells. Fanale MA, et al. reported the results of a phase I study with weekly dosing of brentuximab vedotin in patients with relapsed/refractory CD30-positive hematologic malignancies (Clin Cancer Res. 2012) showed tumor regression in 85% of patients. Thus, the overall objective response rate was 59% (24/44) including 34% (n = 14) of complete remissions. This study mainly included Hodgkin lymphoma (n = 38) and anaplastic large cell lymphoma (n = 5). However, its efficacy in other types of NHL has never been reported although this study enrolled one patient with peripheral T-cell lymphoma not otherwise specified (PTCL-NOS).

CD30 (TNFRSF8) is a transmembrane glycoprotein of the tumor necrosis factor receptor (TNFR) superfamily, and it is involved in signal transduction via the activation of the NF-κB pathway and the mitogen-activated protein kinases (MAPKs), ultimately modulating cell growth, proliferation and apoptosis. CD30 is a non-lineage-specific activation marker expressed by scattered B and T immunoblasts. In addition, a subset of cases in virtually all T-cell lymphoma entities may also express CD30 but at variable and generally lower levels. In fact, a recent study in 22 patients with extranodal NK/T-cell lymphoma showed 75% of positive rate of CD30 expression (75%). Moreover, CD30 expression was also documented in the tumor sample of EB virus positive diffuse large B-cell lymphomas (EBV + DLBCL) of the elderly (28.9%, 11/38). Therefore, Brentuximab vedotin may have potential benefits for patients with CD30-positive NHL other than anaplastic large cell lymphoma such as CD30-positive PTCLs, NOS. Considering the role of CD30 in signal transduction pathway associated with tumor growth and proliferation, its expression may be associated with tumor aggressiveness. In accordance with this, it is more likely that relapse or refractory NHLs may have CD30 expression, and the potential benefits of this promising agent as a salvage therapy deserve to be further investigated in these patients who have high risk of treatment failure. Thus, we designed a phase II study for relapsed or refractory NHL patients. This study is to explore the safety and activity of dosing once every 3 weeks of Brentuximab vedotin in patients with relapsed or refractory CD30-positive NHL other than anaplastic large cell lymphoma.

DETAILED DESCRIPTION:
The principal investigator use a Simon two-stage minimax design based on overall response rates. Overall disease control rates will be calculated as the percent of patients that have confirmed complete response (CR) or partial response (PR) or stable disease (SD) by radiographic response including CT and/or PET scans. We assume a P0 as 20%, and designate a target rate (P1) as 40%. Under the error probabilities (α=0.05, β=0.20), eighteen patients will be enrolled in the first stage. If overall disease control rate is ≤ 4/18 in the first stage, this study will be stopped. If not, this study will recruit patients up to 33 considering 20% of drop out rate.

Intent-to-treat analysis will be applied to all primary and secondary efficacy endpoints. Response rate will be analyzed based on the response criteria according to Cheson 2007 (Cheson BD, et al. J Clin Oncol 2007; 25 (5):579-586), and data related to overall response rate will be analyzed by statistical analysis including Chi test to evaluate predictive factors for response to study drug.

Overall rate of disease control : CR, PR and SD Progression-free survival : Time between the date of treatment start and the date of death due to any cause or date of disease progression (Up to 36months) Data related to survival rate for all patients will be analyzed based on log-rank test by the Kaplan-Meier method.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed non-Hodgkin lymphomas with CD 30 expression. Criteria of positive CD30 expression are defined as in cases with membranous CD30 expression from more than 50% of neoplastic cells.
2. Relapsed or progressed disease after two or more than two salvage chemotherapy
3. Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.
4. Measurable disease > 1.5 cm evidenced by computed tomography (CT) scan of the neck/chest/abdomen/pelvis or CT/positron emission tomography (PET) scans
5. Life expectancy of greater than 3 months
6. ECOG performance status ≤ 2
7. Male or female patients 18 - 75 years
8. Female patient is either post-menopausal for at least 1 year before the screening visit or surgically sterile or if of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 6 months after the last dose of study drug, or agrees to completely abstain from heterosexual intercourse.
9. Male patients, even if surgically sterilized, (i.e., status post vasectomy) agree to practice effective barrier contraception during the entire study period and through 6 months after the last dose of study drug, or agrees to completely abstain from heterosexual intercourse.
10. Voluntary written informed consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
11. Clinical laboratory values as specified below within 7 days before the first dose of study drug:
12. Serum creatinine must be < 2.0 mg/dL and/or creatinine clearance or calculated creatinine clearance > 40 mL/minute.
13. Hemoglobin must be ≥ 8g/dL.
14. Absolute neutrophil count (ANC) ≥ 1500/uL
15. Platelets (Plts) ≥ 75,000/; G-CSF can be given prior to start of brentuximab vedotin and during brentuximab vedotin treatment to achieve target ANC; platelet transfusion can also be given prior to the start of brentuximab vedotin and during brentuximab vedotin treatment to achieve a target platelet ≥ 75,000/uL
16. Total bilirubin within 1.5 x of the upper limit of normal (ULN) institutional limits, patients with elevation of unconjugated bilirubin alone, as in Gilbert's disease, are eligible
17. Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) < 2.5 X institutional ULN. AST and ALT may be elevated up to 5 times the ULN if their elevation can be reasonably ascribed to the presence of hematologic/solid tumor in liver

Exclusion Criteria:

1. Hodgkin lymphoma
2. Anaplastic large cell lymphoma
3. Female patient who are both lactating and breast-feeding or have a positive serum pregnancy test during the screening period or a positive pregnancy test on Day 1 before first dose of study drug
4. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to the protocol.
5. Known cerebral or meningeal disease (HL or any other etiology), including signs or symptoms of PML
6. Symptomatic neurologic disease compromising normal activities of daily living or requiring medications
7. Any sensory or motor peripheral neuropathy greater than or equal to Grade 2
8. Any active systemic viral, bacterial, or fungal infection requiring systemic antibiotics within 2 weeks prior to first study drug dose
9. Any prior treatment with chemotherapy and/or investigational agents completed less than 5 half-lives
10. Known hypersensitivity to recombinant proteins, murine proteins, or to any excipient contained in the drug formulation of brentuximab vedotin.
11. Known HIV antibody-positive
12. Known hepatitis B surface antigen-positive, or known or suspected active hepatitis C infection
13. Diagnosed or treated for another malignancy within 3 years before the first dose or previously diagnosed with another malignancy and have evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
14. Known history of any of the following cardiovascular conditions:

    * Myocardial infarction within 2 years of first dose of study drug
    * New York Heart Association (NYHA) Class III or IV heart failure (see Appendix 3)
    * Evidence of current uncontrolled cardiovascular conditions, including cardiac arrhythmias, congestive heart failure (CHF), angina, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
    * A left-ventricular ejection fraction <50% documented within 6 months before first dose of study drug

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Overall disease control rate | Until the disease progression (maximum 2 years after completion of treatment, assessed up to 36 months)
  The percentage of subjects with complete response (CR) or partial response (PR) or stable disease (SD)

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Time between the date of treatment start and the date of death due to any cause or date of disease progression, whichever came first, assessed up to 36months
Toxicity (assessed by analyzing adverse events and the standard clinical laboratory and hematologic findings.) | From the date of first drug administration until the date of the 30th days, assessed up to 13 months
  Toxicity will be assessed by analyzing adverse events and the standard clinical laboratory and hematologic findings.
Overall survival (OS) | Time between the date of treatment start and the date of death due to any cause,assessed up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Cheolwon Suh, M.D., Principal Investigator — Asan Medical Center; JinSeok Kim, M.D., Principal Investigator — Severance Hospital; HyeonSeok Eom, M.D., Principal Investigator — National Cancer Center of Korea; HyeJin Kang, M.D., Principal Investigator — Korea Cancer Center Hospital
Locations (4):
- South Korea (4):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Yonsei Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Korean Cancer Center Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Kim SJ, Yoon DH, Kim JS, Kang HJ, Lee HW, Eom HS, Hong JY, Cho J, Ko YH, Huh J, Yang WI, Park WS, Lee SS, Suh C, Kim WS. Efficacy of Brentuximab Vedotin in Relapsed or Refractory High-CD30-Expressing Non-Hodgkin Lymphomas: Results of a Multicenter, Open-Labeled Phase II Trial. Cancer Res Treat. 2020 Apr;52(2):374-387. doi: 10.4143/crt.2019.198. Epub 2019 Aug 13. PMID 31476851